CLINICAL TRIAL: NCT03816982
Title: Single-Injection Bupivacaine HCl Plus Either Single-Injection Liposomal Bupivacaine Interscalene Nerve Block or a Continuous Interscalene Nerve Block For Major Shoulder Arthroscopy
Brief Title: Interscalene Bupivacaine With Either Liposomal Bupivacaine or Continuous Peripheral Nerve Block for Shoulder Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Anthony Machi, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU 082018-017
Record Dates: First submitted 2019-01-19; First posted 2019-01-25 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Intervention Model Description: A randomized prospective noninferiority trial to assess the difference, if any, in median pain scores between two block methods using bupivacaine HCl and/or Liposomal bupivacaine, with the catheter method or single shot administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bupivacaine HCl/Bupivacaine CISB (Active Comparator): 23 patients will be enrolled to receive a single-injection bupivacaine HCL interscalene block with bupivacaine CISB added.
  Interventions: Procedure: Single-injection bupivacaine HCl plus a subsequent bupivacaine CISB
- Liposomal Bupivacaine Added to Interscalene Block (Experimental): 23 patients will be enrolled to receive a single-injection bupivacaine HCl interscalene block with liposomal bupivacaine added to same injection.
  Interventions: Procedure: Single-injection bupivacaine HCl plus liposomal bupivacaine

INTERVENTIONS:
Procedure: Single-injection bupivacaine HCl plus liposomal bupivacaine — Patients in the liposomal bupivacaine with added bupivacaine HCl ISB group will be given a single injection LB ISB in the preoperative area only by faculty who are part of the regional anesthesia division. The injectate will include liposomal bupivacaine 10ml (133mg) mixed with bupivacaine HCl 0.5% 10 ml.
  Arms: Liposomal Bupivacaine Added to Interscalene Block
Procedure: Single-injection bupivacaine HCl plus a subsequent bupivacaine CISB — Patients in the bupivacaine CISB group will undergo catheter placement with ultrasound guidance only by faculty who are part of the regional anesthesia division. A 20 mL single bolus ISB with 0.25% bupivacaine will be administered followed by catheter infusion of 0.125% bupivacaine at a rate of 5mL/hour postoperatively by the ON-Q pump
  Arms: Bupivacaine HCl/Bupivacaine CISB

SUMMARY:
This investigation will be a prospective, randomized trial. The study population will consist of adult patients scheduled to undergo major shoulder arthroscopy procedures with anesthesiology at the Ambulatory Services Center (Outpatient Surgery Center). Forty-six subjects will be enrolled in this study and will be randomized into one of two arms: 1) Single-injection bupivacaine HCl plus a subsequent bupivacaine CISB, 2) Single-injection bupivacaine HCl plus liposomal bupivacaine included in the same injection. These procedures will take place, using an ultrasound-guided method, approximately one hour prior to surgical procedure. Subjects will be followed for seven days to assess pain control by the Modified Brief Pain Inventory (MBPI) survey and outcome factors related to study and procedure using the American Shoulder and Elbow Surgeon Shoulder Score (ASES Shoulder Score).

DETAILED DESCRIPTION:
Once potential candidates are identified, charts will be reviewed for initial data collection and to determine if the patient meets inclusion criteria and is free of exclusion criteria. Eligible individuals will be approached in clinic or will be called one to four days before their scheduled procedure and introduced to the study. They will have the opportunity to have the consent and HIPPA forms emailed to them to review before making the decision to participate in the study.

After consent, subjects will be randomized and enrolled into the study. Subjects will be randomized into one of two arms: 1) Single-injection bupivacaine HCl plus a subsequent bupivacaine CISB, 2) Single-injection bupivacaine HCl plus liposomal bupivacaine included in the same injection. Subjects in the first arm will undergo catheter placement with ultrasound guidance by a regional anesthesiologist on the study team. A 20 mL single bolus ISB with 0.25% bupivacaine will be administered followed by catheter infusion of 0.125% bupivacaine at a rate of 5 mL/hour postoperatively by the elastomeric pump. Subjects in the second arm will be given a single injection Liposomal Bupivacaine ISB in the preoperative area by a regional anesthesiologist on the study team. The injectate will include liposomal bupivacaine 10 mL (133 mg) mixed with bupivacaine HCl 0.5% 10 mL.

Both groups will receive a standardized analgesic regimen which will include the following: preoperative acetaminophen 15mg/kg up to 1gm PO and gabapentin 600 mg PO; intraoperative dexamethasone 8mg IV, fentanyl 100 - 250 mcg IV, ketamine 30 -50mg IV, and ketorolac 0.5mg/kg up to 30mg IV at conclusion of surgery; fentanyl IV in PACU as necessary; postoperative regimen will include acetaminophen 15mg/kg up to 1gm PO q8hrs, ibuprofen 400 mg Q8 hrs and tramadol 50 mg q4hrs prn. For continued breakthrough postoperative pain unrelieved adequately by tramadol a patient may receive oxycodone 5mg PO every 4 hours as needed.

Subjects in both groups will receive baseline ASES Shoulder Score assessments before the block and procedure, and again in postoperative days 1-7. Additionally, a daily MBPI Short Form will be adminstered for the seven days post operation. The primary endpoint is to assess the median pain score on POD 1 using the MBPI Short form. Secondary endpoints include Cumulative Area Under Curve (AUC) median pain score on POD1-3, opioid consumption through POD3, satisfaction with pain treatment, block duration, success rate, amount of analgesia/sedation used for it; and adverse effects attributed to either the block or catheter, and functionality of the surgical arm.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years
* Individuals presenting for major shoulder arthroscopy procedures at Ambulatory Services Center (Outpatient Surgery Center) -that include rotator cuff repair and biceps tenodesis
* Patient is able to provide informed consent to participate in the study.

Exclusion Criteria:

* Allergy to amide local anesthetic, liposomal bupivacaine or other medication involving liposomal formulation
* Preexisting neurological deficits involving or potentially involving the ipsilateral brachial plexus
* Preexisting contralateral vocal fold paralysis or recurrent laryngeal paralysis
* Psychiatric or cognitive disorders that could interfere with perioperative evaluation including drug or alcohol abuse
* Chronic pain conditions
* Preoperative opioid consumption greater than 20 mg oral morphine equivalent.
* Any contraindication to interscalene nerve block including any local disorder of the skin where blockade is to be performed which would prevent safe performance of the block
* Any coagulation abnormality which would be a contraindication for block placement
* Preoperative chronic renal dysfunction requiring renal replacement therapy or a serum creatinine greater than 1.4 mg/dL
* Body mass index >50
* Pregnancy
* Incarceration
* ASA classification greater than 3
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Median pain score on POD1 | 24 hours
  Median pain score on POD1 as measured by the MBPI Short Form

SECONDARY OUTCOMES:
Cumulative Area under Curve median pain score on POD1-3 | 72 hours
  Median pain score on POD1-3 as measured by the MBPI Short Form

CONTACTS AND LOCATIONS:
Overall Officials: Anthony T Machi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No study data will be shared with outside entities or non-IRB approved study personnel.